CLINICAL TRIAL: NCT03266172
Title: A Three Part, Non-randomized, Open Label Study Designed to Assess the Pharmacokinetics of GSK2982772 Following Administration of Minitab Modified Release Formulations in a Capsule Relative to an Immediate Release Reference Tablet Formulation (Part A), the Pharmacokinetics of Escalating, Repeat Doses of a Selected Minitab Modified Release Prototype (Part B) , and the Pharmacokinetics of GSK2982772 Following Administration of Modified Release Tablet Formulations in the Fed and Fasted State (Part C) in Healthy Participants
Brief Title: A Study to Compare the Pharmacokinetics (PK) of GSK2982772 Following Administration of Different Modified Release (MR) Formulations in Capsule and MR Tablet Formulations Relative to an Immediate Release (IR) Tablet Formulation and to Check the PK of MR Formulation in Capsule Following Repeat Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 205017
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Results first posted 2020-01-09 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Autoimmune Diseases
Keywords: immediate release tablet; GSK2982772; Modified release; minitablet
MeSH Terms: conditions — Autoimmune Diseases | interventions — GSK2982772

STUDY DESIGN:
Intervention Model Description: Part A of the study will be a non-randomized 6 period, sequential, 6-way fixed sequence design. Part B of the study will be a repeat dose study. Part C of the study will be a non-randomized 6 period, sequential, fixed sequence crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjects in Part A (Experimental): Subjects in Part A will receive GSK2982772 MR (Period 1, 2, 4, 5 and 6) and GSK2982772 IR (Period 3)
  Interventions: Drug: GSK2982772 Modified Release; Drug: GSK2982772 Immediate Release
- Subjects in Part B (Experimental): Subjects in Part B will receive GSK2982772 MR
  Interventions: Drug: GSK2982772 Modified Release
- Subjects in Part C (Experimental): Subjects in Part C will receive GSK2982772 MR (Period 1, 3, 4, 5 and 6) and GSK2982772 IR (Period 2)
  Interventions: Drug: GSK2982772 Modified Release; Drug: GSK2982772 Immediate Release

INTERVENTIONS:
Drug: GSK2982772 Modified Release — GSK2982772 MR will be available as prototype MR minitablet in capsules with unit dose strength of 60 mg in Part A. In Part B, GSK2982772 MR minitablet in capsules with unit dose strength of 15, 30 or 60 mg will be administered by subjects for Days 1 to 3. In Part C, GSK2982772 MR tablet with unit dose strength of 240, 360 or 480 mg will be administered by subjects. GSK2982772 MR will be administered orally with 240 mL of water.
Drug: GSK2982772 Immediate Release — In part A, GSK2982772 IR tablet will be available with unit dose strength of 30 mg and the total dose administered by subjects will be 120 mg (4 tablets of dose strength 30 mg) orally with 240 mL of water. In part C, GSK2982772 IR tablet will be available with unit dose strength of 30 mg and the total dose administered by subjects will be 240 mg (8 tablets of dose strength 30 mg) orally with 240 mL of water.
  Arms: Subjects in Part A; Subjects in Part C

SUMMARY:
GSK2982772 is a first-in-class, highly selective, receptor-interacting protein-1 (RIP1) kinase inhibitor being developed for the treatment of inflammatory bowel disease, plaque psoriasis (PsO), rheumatoid arthritis (RA) and other disease conditions. PK data from the first time in human (FTIH) study for GSK2982772 showed that the half life of GSK2982772 was short (approximately 2 to 3 hours). A once daily (QD) formulation would be more convenient from a subject perspective and could offer the advantage of providing a flatter GSK2982772 concentration time profile. Following completion of Parts A and B, it was determined that the slowest minitab formulation provided a PK profile suitable for QD dosing but this formulation was susceptible to a food effect. This study will evaluate the pharmacokinetics of GSK2982772 following administration of different minitab MR formulations in a capsule relative to an IR reference tablet formulation, the pharmacokinetics of selected MR formulation in capsule following repeat doses for 3 days and to compare the pharmacokinetics of GSK2982772 following administration of MR tablet formulations in the fed and fasted state relative to an IR tablet formulation. The study is divided into three parts: Part A will be a non-randomized 6 periods, sequential, 6-way fixed sequence design in which up to 4 MR minitab formulations in a capsule will be evaluated. Periods 1, 2, and 3 will evaluate a slow MR release duration (nominally 24 hours), a fast MR release duration (nominally 10 hours), and IR tablet respectively. Periods 4, 5 and 6 will have flexible dose regimen and it will depend on the outcomes of Period 1 to 3. Subjects will be admitted to the clinic the previous day before dosing. Each in-patient period will consist of 3 days and 2 nights followed by a minimum washout period of 7 days between doses, for both Part A and C. In Part A and C, 16 healthy subjects will be enrolled such that at least 12 evaluable subjects complete the study. Part B will be an open-label, repeat dose study in which the selected MR minitab formulation in capsule will be evaluated. Each in-patient period will consist of 5 days and 4 nights. There will be a minimum of 7 days washout period between the last morning dose of one period and the first dose of the next period. In Part B, 10 healthy subjects will be enrolled such that at least 6 evaluable subjects complete the study. Part C of the study will be a non-randomised 6 period, sequential, fixed sequence crossover design in which MR tablet formulations will be evaluated. Periods 1 and 2 will evaluate single dose administration of a 240 milligram (mg) MR tablet and the 240 mg IR tablet (reference), respectively. Periods 3, 4, 5 and 6 will be flexible and the dosing regimen will be dependent on the outcome of Periods 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body weight greater than and equal to 50 kilogram (kg) and body mass index within the range 19.0 to 32.0 kilogram per meter square (kg/m^2) (inclusive).
* A male subject must agree to use a highly effective contraception during the treatment period and for at least 90 days after the last dose of study treatment and refrain from donating sperm during this period.
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive during the treatment period and for at least 30 days before and 30 days after the last dose of study treatment.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Parts A and C only: Any history of suicidal behavior within the past 6 months or any history of attempted suicide in a subject's lifetime.
* Part B only: Subjects with current history of suicidal ideation behavior as measured using the columbia-suicide severity rating scale (C-SSRS) or a history of attempted suicide.
* History of clinically significant psychiatric disorders as judged by the investigator. Depression requiring treatment in the last 2 years.
* History of herpes zoster (shingles) reactivation.
* History or diagnosis of obstructive sleep apnea.
* History of a significant respiratory disorder. Childhood asthma that has fully resolved is permitted.
* History or current evidence of febrile seizures, epilepsy, convulsions, significant head injury, or other significant neurologic conditions.
* A positive diagnostic tuberculosis (TB) test at screening defined as a positive QuantiFERON-TB Gold test or T-spot test. In cases where the QuantiFERON or T spot test is indeterminate, the subject may have the test repeated once, but they will not be eligible for the study unless the second test is negative.
* History of GI surgery (with exception of appendectomy).
* History of cholecystectomy or gall stones.
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active.
* ALT greater than 1.5 times upper limit of normal (ULN).
* Bilirubin greater than 1.5 times ULN (isolated bilirubin greater than 1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35 percentage of total).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome).
* Corrected QT interval (QTc) greater than 450 millisecond (msec).
* Past or intended use of over-the-counter or prescription medication including herbal medications within 7 days prior to dosing (paracetamol/acetaminophen [up to 2 gram (g) per day], hormone replacement therapy and hormonal contraception are permitted).
* Live or attenuated vaccine(s) within 30 days of enrolment, or plans to receive such vaccines during the study or plans to receive a vaccine within 30 days + 5 half-lives of the last dose of study medication.
* Subject in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within a 56 day period; therefore donation or loss of greater than 400 mL of blood within the previous 3 months.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation within the last 3 months before signing of consent in this or any other clinical study involving an investigational study treatment or any other type of medical research.
* Subjects who have previously been enrolled in this study. Subjects in Part A of this study are not permitted to participate in Part B. Subjects in Parts A or B of this study are not permitted to participate in Part C.
* Current or history of renal disease or estimated glomerular filtration rate (GFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation calculation less than 60 mL/minutes(min)/1.73m^2 at screening.
* Presence of Hepatitis B surface antigen (HBsAg) at screening Positive Hepatitis C antibody test result at screening or within 3 months prior to first dose. As potential for and magnitude of immunosuppression with this compound is unknown, subjects with presence of hepatitis B core antibody (HBcAb) should be excluded. Subjects positive for HBsAg and/or positive for anti-HBc antibody (regardless of anti-HBs antibody status) are excluded.
* An elevated C-reactive protein (CRP) outside the normal reference range.
* Part B only: A positive anti-nuclear antibody (ANA) outside the normal reference range.
* Confirmed positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse, or history of drug or alcohol abuse in the past 5 years.
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of greater than 21 units for males or greater than 14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Current use or history of regular use of tobacco- or nicotine-containing products within 6 months prior to screening. A carbon monoxide breath test reading of greater than 10 parts per million (ppm).
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Unwilling or unable to swallow multiple size 0-00 capsules as part of study participation.
* Subjects who do not have suitable veins for multiple venipunctures/cannulation as assessed by the investigator at screening.
* Total cholesterol greater than or equal to 300 milligram/deciliter (mg/dL) (greater than or equal to 7.77 millimoles per liter [mmol]/L]) or triglycerides greater than or equal to 250 mg/dL (greater than or equal to 2.82 mmol/L).
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20863

REFERENCES:
- [Background] Tompson DJ, Whitaker M, Pan R, Johnson G, Fuller T, McKenzie L, Zann V, Powell M, Abbott-Banner K, Hawkins S. Development of a Prototype, Once-Daily, Modified-Release Formulation for the Short Half-Life RIPK1 Inhibitor GSK2982772. Pharm Res. 2021 Jul;38(7):1235-1245. doi: 10.1007/s11095-021-03059-z. Epub 2021 Jun 16. PMID 34136987

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, 3-part, single and repeat dose study conducted in healthy participants to assess modified release (MR) minitablets (MT) in a capsule and MR monolithic matrix (MM) formulations of GSK2982772 compared to immediate release (IR) tablet formulation of GSK2982772.
Pre-assignment Details: In this study, total 45 participants were enrolled.
Groups:
- MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat): Participants in Part A received a single dose of 120 mg GSK2982772 MR MT-12hour (hr) capsule (80% release at 12 hours) in fasted state in Period 1 followed by a single dose of 120 mg GSK2982772 MR MT-8hour capsule (80% release at 8 hours) in fasted state in Period 2. In Period 3, participants received a single oral dose of 120 milligram (mg) GSK2982772 (4x30 mg) IR tablet in fasted state followed by a single oral dose of 120 mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) after high fat meal in Period 4. There was a washout period of 7 days between each treatment period. All doses were administered via the oral route with 240 milliliters (mL) of water.
- MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard): Participants in Part B received once daily dose of 120mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fasted state for 3 days in Period 1 followed by once daily dose of 240mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fasted state for 3 days in Period 2. In Period 3, participants received once daily dose of 300mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fed state (standard meal) for 3 days. There was washout period of 7 days between each treatment period. All doses were administered via oral route with 240 mL water.
- MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF: Participants in Part C received a single dose of 240 mg GSK2982772 MR MM-12hour tablet (80% release at 12 hours) in fasted (Fast) state in Period 1 followed by a single dose of 240 mg GSK2982772 IR tablet in fasted state in Period 2. In Period 3, participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fasted state. In Period 4, participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fed state followed by a single dose of 480 mg GSK2982772 MR MM-12hours (80% release at 12 hours) before standard breakfast (delayed fed [DF]) in Period 5. In Period 6, participants received a single dose of 240 mg GSK2982772 MR MM-12hours (80% release at 12 hours) before high-fat breakfast (DF). There was a washout period of 7 days between each treatment period. All doses were administered via oral route with 240 mL water
Period: Part A: Period 1(2 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 16 | 0 | 0
Completed | 15 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Part A: Washout Period (7 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 15 | 0 | 0
Completed | 13 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Part A: Period 2 (2 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 13 | 0 | 0
Completed | 13 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part A: Washout (7 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 13 | 0 | 0
Completed | 13 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part A: Period 3 (2 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 16 (3 replacement participants were enrolled) | 0 | 0
Completed | 16 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part A: Washout (7 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 16 | 0 | 0
Completed | 16 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part A: Period 4 (2 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 16 | 0 | 0
Completed | 16 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part B: Period 1 (4 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 (Participants from Part A did not enter Part B) | 10 (New participants were enrolled in Part B of study) | 0
Completed | 0 | 10 | 0
Not Completed | 0 | 0 | 0
Period: Part B: Washout (7 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 10 | 0
Completed | 0 | 10 | 0
Not Completed | 0 | 0 | 0
Period: Part B: Period 2 (4 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 10 | 0
Completed | 0 | 10 | 0
Not Completed | 0 | 0 | 0
Period: Part B: Washout (7 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 10 | 0
Completed | 0 | 8 | 0
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Period: Part B: Period 3 (4 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 6 (Two participants completed Washout Period but withdrew before the start of Period 3.) | 0
Completed | 0 | 6 | 0
Not Completed | 0 | 0 | 0
Period: Part C: Period 1(2 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 0 (Participants from Part B did not enter Part C) | 15 (New participants were enrolled in Part C of study)
Completed | 0 | 0 | 15
Not Completed | 0 | 0 | 0
Period: Part C Washout Period (7 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 0 | 15
Completed | 0 | 0 | 15
Not Completed | 0 | 0 | 0
Period: Part C Period 2(2 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 0 | 15
Completed | 0 | 0 | 15
Not Completed | 0 | 0 | 0
Period: Part C Washout Period (7 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 0 | 15
Completed | 0 | 0 | 15
Not Completed | 0 | 0 | 0
Period: Part C Period 3(2 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 0 | 16 (1 replacement participant enrolled)
Completed | 0 | 0 | 16
Not Completed | 0 | 0 | 0
Period: Part C Washout Period (7 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 0 | 16
Completed | 0 | 0 | 16
Not Completed | 0 | 0 | 0
Period: Part C Period 4(2 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 0 | 16
Completed | 0 | 0 | 16
Not Completed | 0 | 0 | 0
Period: Part C Washout Period (7 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 0 | 16
Completed | 0 | 0 | 15
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Part C Period 5(2 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 0 | 15
Completed | 0 | 0 | 15
Not Completed | 0 | 0 | 0
Period: Part C Washout Period (7 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 0 | 15
Completed | 0 | 0 | 14
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Part C Period 6(2 Days)
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF
Started | 0 | 0 | 14
Completed | 0 | 0 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF: Participants in Part C received a single dose of 240 mg GSK2982772 MR MM-12hour tablet (80% release at 12 hours) in fasted (Fast) state in Period 1 followed by a single dose of 240 mg GSK2982772 IR tablet in fasted state in Period 2. In Period 3, participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fasted state. In Period 4, participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fed state followed by a single dose of 480 mg GSK2982772 MR MM-12hours (80% release at 12 hours) before standard breakfast (delayed fed [DF]) in Period 5. In Period 6, participants received a single dose of 240 mg GSK2982772 MR MM-12hours (80% release at 12 hours) before high-fat breakfast (delayed fed). There was a washout period of 7 days between each treatment period. All doses were administered via oral route with 240 mL water
- Total: Total of all reporting groups
Arm/Group | MT-12hr Fasted/MT-8hr Fasted/IR Fasted/MT-12hr Fed (High Fat) | MT 120mg Fasted/MT 240mg Fasted/ MT 300mg Fed (Standard) | MM240 Fast/IR240 Fast/MM480 Fast/MM480 Fed/MM480 DF/MM240 DF | Total
Number analyzed (Participants) | 19 | 10 | 16 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (14.10) | 47.8 (13.43) | 45.3 (12.22) | 47.5 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 7 | 19
  Male | 11 | 6 | 9 | 26
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 1 | 0 | 1 | 2
  White - White/Caucasian/European Heritage | 18 | 10 | 14 | 42
  Asian - South East Asian Heritage | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Infinity (AUC[0-inf]) of GSK2982772 in IR Formulation: Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-inf). Participants in the 'Safety Population' for whom a Pharmacokinetic (PK) sample was obtained and analyzed were part of PK Population.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part A: IR 120mg Fasted: Participants received a single oral dose of 120 mg GSK2982772 (4x30 mg) IR tablet in fasted state
Arm/Group | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16
Hours*microgram per milliliter | 6.305 (39.4)

2. Primary Outcome: AUC(0-inf) of GSK2982772 in MT Formulation :Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-inf).
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population. Only those participants with data available at specified time frame were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part A: MT-12hour 120mg Fasted: Participants received a single dose of 120 mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fasted state
- Part A: MT-8hour 120mg Fasted: Participants received single dose of 120 mg GSK2982772 MR MT-8hour capsule (80% release at 8 hours) in fasted state
- Part A: MT-12hour 120mg Fed (High Fat): Participants received single oral dose of 120 mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) after high fat meal
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 10 | 10 | 10
Hours*microgram per milliliter | 3.852 (39.4) | 4.482 (47.4) | 5.314 (39.7)

3. Primary Outcome: Area Under the Curve From Time Zero to the Last Measurable Concentration (AUC[0-t]) of GSK2982772 in IR Formulation : Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-t)
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16
Hours*microgram per milliliter | 6.258 (39.2)

4. Primary Outcome: AUC(0-t) of GSK2982772 in MT Formulation: Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-t)
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population. Only those participants with data available at specified time frame were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part A:MT-8hour 120mg Fasted: Participants received single dose of 120 mg GSK2982772 MR MT-8hour capsule (80% release at 8 hours) in fasted state
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A:MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 13 | 15
Hours*microgram per milliliter | 3.805 (42.3) | 4.449 (49.4) | 4.720 (38.4)

5. Primary Outcome: Area Under the Curve From Time Zero to 24 Hours (AUC[0-24]) of GSK2982772 in IR Formulation: Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-24)
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16
Hours*microgram per milliliter | 6.256 (39.2)

6. Primary Outcome: AUC(0-24) of GSK2982772 in MT Formulation: Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-24)
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population. Only those participants with data available at specified time frame were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part A:MT-12hour 120mg Fasted: Participants received a single dose of 120 mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fasted state
Arm/Group | Part A:MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 13 | 15
Hours*microgram per milliliter | 3.558 (43.6) | 4.255 (49.4) | 4.580 (39.5)

7. Primary Outcome: Area Under the Curve From Time Zero to 12 Hours (AUC[0-12]) of GSK2982772 in IR Formulation: Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-12)
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16
Hours*microgram per milliliter | 5.967 (38.4)

8. Primary Outcome: AUC(0-12) of GSK2982772 in MT Formulation: Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-12)
Time Frame: Pre-dose, 2, 4, 6, 8, 10, and 12 hours post-dose
Population: PK Population. Only participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part A:MT-12hour 120mg Fasted | Part A:MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 13 | 15
Hours*microgram per milliliter | 2.106 (45.1) | 3.066 (47.7) | 3.573 (40.8)

9. Primary Outcome: Maximum Observed Concentration (Cmax) of GSK2982772 in IR Formulation: Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for Cmax
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16
Microgram per milliliter | 1.375 (40.1)

10. Primary Outcome: Cmax of GSK2982772 in MT Formulation: Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for Cmax
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population. Only participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 13 | 15
Microgram per milliliter | 0.277 (58.8) | 0.439 (54.9) | 0.624 (49.4)

11. Primary Outcome: Concentration at 12 Hours Post-dose (C12hour) of GSK2982772 in Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for C12hour.
Time Frame: 12 hours post-dose
Population: PK Population. Only participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat) | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16 | 13 | 15 | 16
Microgram per milliliter | 0.220 (52.6) | 0.209 (56.2) | 0.208 (53.1) | 0.045 (81.7)

12. Primary Outcome: Concentration at 24 Hours Post-dose (C24hour) of GSK2982772 in Part A
Description: Blood samples were collected from participants at indicated time points and analyzed for C24hour.
Time Frame: 24 hours post-dose
Population: PK Population. Only participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat) | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16 | 13 | 15 | 16
Microgram per milliliter | 0.058 (73.2) | 0.046 (69.5) | 0.030 (46.6) | 0.006 (108.8)

13. Primary Outcome: Relative Bioavailability (Frelformulation) Based on AUC (0-inf) of GSK2982772 in Part A
Description: Blood samples were collected at indicated time points for analysis of Frelformulation. Frelformulation for AUC (0-inf) was calculated as Geometric mean of AUC (0-inf) of MT (test) / Geometric mean of AUC (0-inf) of IR Formulation (reference) multiplied by 100.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose (reference); Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 26, 28, 30 and 32 hours post-dose (test)
Population: PK Population. Only those participants with data available at specified time frame were analyzed.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Groups:
- Part A:120 mg MT-8hr Fasted and 120 mg IR Fasted: Participants received single dose of 120 mg GSK2982772 MR MT-8hour capsule (80% release at 8 hours) in fasted state and received single oral dose of 120 mg GSK2982772 (4x30 mg) IR tablet in fasted state. There was washout period of 7 days between doses
- Part A:120 mg MT-12hr Fasted and 120 mg IR Fasted: Participants received a single dose of 120 mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fasted state and received single oral dose of 120 mg GSK2982772 (4x30 mg) IR tablet in fasted state. There was washout period of 7 days between doses
Arm/Group | Part A:120 mg MT-8hr Fasted and 120 mg IR Fasted | Part A:120 mg MT-12hr Fasted and 120 mg IR Fasted
Number analyzed (Participants) | 10 | 10
Percentage bioavailability | 72.77 [67.91 to 77.98] | 60.53 [56.15 to 65.24]

14. Primary Outcome: Frelformulation Based on AUC (0-24) of GSK2982772 in Part A
Description: Blood samples were collected at indicated time points for analysis of Frelformulation. Frelformulation for AUC (0-24) was calculated as Geometric mean of AUC (0-24) of MT (test) / Geometric mean of AUC (0-24) of IR Formulation (reference) multiplied by 100.
Time Frame: Pre-dose 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose (reference); Pre-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 24 hours post-dose (test)
Population: PK Population. Only those participants with data available at specified time frame were analyzed.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part A:120 mg MT-8hr Fasted and 120 mg IR Fasted | Part A:120 mg MT-12hr Fasted and 120 mg IR Fasted
Number analyzed (Participants) | 13 | 16
Percentage bioavailability | 68.18 [63.98 to 72.64] | 57.54 [54.01 to 61.30]

15. Primary Outcome: Frelformulation Based on Cmax of GSK2982772 in Part A
Description: Blood samples were collected at indicated time points for analysis of Frelformulation. Frel was calculated as Geometric mean of Cmax of MT Formulation (test)/ Geometric mean of Cmax of IR Formulation (reference) multiplied by 100.
Time Frame: Pre-dose,0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose(reference); Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 26, 28, 30 and 32 hours post-dose(test)
Population: PK Population. Only those participants with data available at specified time frame were analyzed.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part A:120 mg MT-8hr Fasted and 120 mg IR Fasted | Part A:120 mg MT-12hr Fasted and 120 mg IR Fasted
Number analyzed (Participants) | 13 | 16
Percentage bioavailability | 32.13 [27.36 to 37.75] | 20.39 [17.41 to 23.89]

16. Primary Outcome: Ratio of Cmax to C12hour of GSK2982772 in IR Formulation: Part A
Description: Blood samples were collected at indicated time points for analysis of ratio of Cmax to C12hour. Mean and standard deviation of ratio of Cmax to C12 hour has been presented.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16
Ratio | 36.485 (20.9265)

17. Primary Outcome: Ratio of Cmax to C12hour of GSK2982772 in MT Formulation: Part A
Description: as for outcome 16
Time Frame: Pre-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population. Only participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 13 | 15
Ratio | 1.284 (0.2468) | 2.265 (0.9119) | 3.240 (1.2250)

18. Primary Outcome: Ratio of Cmax to C24hour of GSK2982772 in IR Formulation: Part A
Description: Blood samples were collected at indicated time points for analysis of ratio of Cmax to C24hour. Mean and standard deviation of ratio of Cmax to C24 hour has been presented.
Time Frame: Pre-dose 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16
Ratio | 312.851 (221.7640)

19. Primary Outcome: Ratio of Cmax to C24hour of GSK2982772 in MT Formulation: Part A
Description: as for outcome 18
Time Frame: Pre-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population. Only participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 13 | 15
Ratio | 6.119 (5.1507) | 10.790 (4.9019) | 22.915 (11.7978)

20. Primary Outcome: Time to Cmax (Tmax) of GSK2982772 in IR Formulation: Part A
Description: Blood samples were collected at indicated time points for analysis of Tmax.
Time Frame: Pre-dose 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16
Hours | 2.000 [0.67 to 3.00]

21. Primary Outcome: Tmax of GSK2982772 in MT Formulation: Part A
Description: Blood samples were collected at indicated time points for analysis of Tmax.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population. Only participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 13 | 15
Hours | 10.000 [2.08 to 18.00] | 4.000 [4.00 to 10.00] | 6.000 [4.00 to 10.00]

22. Primary Outcome: AUC(0-inf) of GSK2982772 for IR Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of AUC (0-inf)
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part C: IR 240mg Fasted: Participants received a single dose of 240 mg GSK2982772 IR tablet in fasted state
Arm/Group | Part C: IR 240mg Fasted
Number analyzed (Participants) | 14
Hours*microgram per milliliter | 14.797 (26.3)

23. Primary Outcome: AUC(0-inf) of GSK2982772 for MM Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of AUC (0-inf).
Time Frame: Pre-dose, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part C: MM-12h 240mg Fasted: Participants received a single dose of 240 mg GSK2982772 MR MM-12hour tablet (80% release at 12 hours) in fasted state
- Part C: MM-12h 480mg Fasted: Participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fasted state
Arm/Group | Part C: MM-12h 240mg Fasted | Part C: MM-12h 480mg Fasted
Number analyzed (Participants) | 4 | 4
Hours*microgram per milliliter | 13.417 (23.4) | 22.493 (51.3)

24. Primary Outcome: AUC(0-t) of GSK2982772 for IR Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of AUC (0-t).
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at specified time frame were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part C: IR 240mg Fasted
Number analyzed (Participants) | 15
Hours*microgram per milliliter | 14.621 (25.7)

25. Primary Outcome: AUC(0-t) of GSK2982772 for MM Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of AUC (0-t).
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part C: MM-12h 240mg Fasted | Part C: MM-12h 480mg Fasted
Number analyzed (Participants) | 15 | 16
Hours*microgram per milliliter | 9.676 (29.6) | 20.009 (29.7)

26. Primary Outcome: AUC(0-24) of GSK2982772 for IR Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of AUC (0-24)
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part C: IR 240mg Fasted
Number analyzed (Participants) | 15
Hours*microgram per milliliter | 14.619 (25.7)

27. Primary Outcome: AUC(0-24) of GSK2982772 for MM Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of AUC (0-24)
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part C: MM-12h 240mg Fasted | Part C: MM-12h 480mg Fasted
Number analyzed (Participants) | 15 | 16
Hours*microgram per milliliter | 8.769 (30.9) | 18.177 (31.5)

28. Primary Outcome: AUC (0-12) of GSK2982772 for IR Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of AUC (0-12)
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part C: IR 240mg Fasted
Number analyzed (Participants) | 15
Hours*microgram per milliliter | 13.500 (26.3)

29. Primary Outcome: AUC (0-12) of GSK2982772 for MM Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of AUC (0-12)
Time Frame: Pre-dose, 2, 4, 6, 8, 10, and 12 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part C: MM-12h 240mg Fasted | Part C: MM-12h 480mg Fasted
Number analyzed (Participants) | 15 | 16
Hours*microgram per milliliter | 6.096 (32.8) | 12.508 (40.1)

30. Primary Outcome: Cmax of GSK2982772 for IR Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of Cmax
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part C: IR 240mg Fasted
Number analyzed (Participants) | 15
Microgram per milliliter | 2.938 (25.2)

31. Primary Outcome: Cmax of GSK2982772 for MM Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of Cmax
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part C: MM-12h 240mg Fasted | Part C: MM-12h 480mg Fasted
Number analyzed (Participants) | 15 | 16
Microgram per milliliter | 0.918 (34.2) | 2.010 (50.1)

32. Primary Outcome: C12 of GSK2982772 in Part C: Fasted State
Description: Blood samples was collected at indicated time point for analysis of C12
Time Frame: 12 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part C: IR 240mg Fasted | Part C: MM-12h 240mg Fasted | Part C: MM-12h 480mg Fasted
Number analyzed (Participants) | 15 | 15 | 16
Microgram per milliliter | 0.197 (62.9) | 0.346 (41.7) | 0.671 (42.3)

33. Primary Outcome: C24 of GSK2982772 in Part C: Fasted State
Description: Blood samples was collected at indicated time point for analysis of C24
Time Frame: 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part C: IR 240mg Fasted | Part C: MM-12h 240mg Fasted | Part C: MM-12h 480mg Fasted
Number analyzed (Participants) | 15 | 15 | 16
Microgram per milliliter | 0.025 (54.9) | 0.162 (52.6) | 0.351 (52.5)

34. Primary Outcome: Ratio of Cmax to C12hour of GSK2982772 for IR Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of ratio of Cmax to C12hour. Mean and standard deviation of ratio of Cmax to C12 hours has been presented.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part C: IR 240mg Fasted
Number analyzed (Participants) | 15
Ratio | 17.158 (7.9158)

35. Primary Outcome: Ratio of Cmax to C12hour of GSK2982772 for MM Formulation in Part C: Fasted State
Description: as for outcome 34
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part C: MM-12h 240mg Fasted | Part C: MM-12h 480mg Fasted
Number analyzed (Participants) | 15 | 16
Ratio | 2.892 (1.2572) | 3.551 (2.2615)

36. Primary Outcome: Ratio of Cmax to C24hour of GSK2982772 for IR Formulation in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of ratio of Cmax to C24hour. Mean and standard deviation of ratio of Cmax to C24 hours has been presented.
Time Frame: Pre-dose,0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part C: IR 240mg Fasted
Number analyzed (Participants) | 15
Ratio | 138.239 (76.3996)

37. Primary Outcome: Ratio of Cmax to C24hour of GSK2982772 for MM Formulation in Part C: Fasted State
Description: as for outcome 36
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part C: MM-12h 240mg Fasted | Part C: MM-12h 480mg Fasted
Number analyzed (Participants) | 15 | 16
Ratio | 6.026 (2.1936) | 7.991 (10.6319)

38. Primary Outcome: Frelformulation Based on AUC (0-t) of GSK2982772 in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of Frelformulation. Frel for AUC (0-t) was calculated as Geometric mean of AUC (0-t) of MM formulation (test) / Geometric mean of AUC (0-t) of IR Formulation (reference) multiplied by 100.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose(reference); Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours post-dose(test)
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Groups:
- Part C:MM-12h 240mg Fasted and IR 240mg Fasted: Participants in received a single dose of 240 mg GSK2982772 MR MM-12hour tablet (80% release at 12 hours) in fasted state and a single dose of 240 mg GSK2982772 IR tablet in fasted state. There was washout period of 7 days between doses
Arm/Group | Part C:MM-12h 240mg Fasted and IR 240mg Fasted
Number analyzed (Participants) | 15
Percentage bioavailability | 66.18 [61.91 to 70.74]

39. Primary Outcome: Frelformulation Based on AUC (0-24) of GSK2982772 in Part C: Fasted State
Description: Blood samples were collected at indicated time points for analysis of Frelformulation. Frel for AUC (0-24) was calculated as Geometric mean of AUC (0-24) of MM Fasted formulation (test) / Geometric mean of AUC (0-24) of IR Formulation (reference) multiplied by 100.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose(reference); Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 hours post-dose(test)
Population: PK Population. Only those participants with data available at the specified data points were analyzed
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part C:MM-12h 240mg Fasted and IR 240mg Fasted
Number analyzed (Participants) | 15
Percentage bioavailability | 59.98 [55.06 to 65.34]

40. Secondary Outcome: Frelformulation Based on AUC (0-inf) of GSK2982772 After a High Fat Meal in Part A
Description: Blood samples were collected at indicated time points for analysis of Frelformulation based on AUC of GSK2982772 after a high fat meal. Frel for AUC (0-inf) was calculated as Geometric mean of AUC (0-inf) of MT Fed formulation (test) / Geometric mean of AUC (0-inf) of MT Fasted Formulation (reference) multiplied by 100.
Time Frame: Pre-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Groups:
- Part A:120 mg MT-12hour Fed and 120 mg MT-12hour Fasted: Participants received single oral dose of 120 mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) after high fat meal and received a single dose of 120 mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fasted state. There was washout period of 7 days between doses
Arm/Group | Part A:120 mg MT-12hour Fed and 120 mg MT-12hour Fasted
Number analyzed (Participants) | 10
Percentage bioavailability | 123.64 [115.98 to 131.80]

41. Secondary Outcome: Frelformulation Based on Cmax of GSK2982772 After a High Fat Meal in Part A
Description: Blood samples were collected at indicated time points for analysis of FrelFE based on AUC of GSK2982772 after a high fat meal. Frel for Cmax was calculated as Geometric mean of Cmax of MT Fed formulation (test) / Geometric mean of Cmax of MT Fasted Formulation (reference) multiplied by 100.
Time Frame: Pre-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population. Only those participants with data available at specified timepoint were analyzed
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part A:120 mg MT-12hour Fed and 120 mg MT-12hour Fasted
Number analyzed (Participants) | 15
Percentage bioavailability | 225.07 [201.78 to 251.04]

42. Secondary Outcome: AUC(0-24) of GSK2982772 in Part B
Description: Blood samples were collected at indicated time points for analysis of AUC (0-24)
Time Frame: Pre-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 hours on Day 1 and Day 3
Population: PK Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram/milliliter
Groups:
- Part B: MT-12 120mg Fasted: Participants received once daily dose of 120mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fasted state for 3 days.
- Part B :MT-12 240mg Fasted: Participants received once daily dose of 240mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fasted state for 3 days
- Part B :MT-12hour 300mg Fed (Standard): Participants received once daily dose of 300mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fed state (standard meal) for 3 days
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Hours*microgram/milliliter
  Day 1, n=10, 9, 5: number analyzed (Participants) | 10 | 9 | 5
  Day 1, n=10, 9, 5 | 4.669 (26.5) | 8.807 (34.3) | 9.662 (33.8)
  Day 3, n=10, 10, 6 | 5.010 (32.0) | 9.867 (30.4) | 10.948 (37.7)

43. Secondary Outcome: Cmax of GSK2982772 in Part B
Description: Blood samples were collected at indicated time points for analysis of Cmax
Time Frame: Pre-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 hours on Day 1 and Day 3
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/milliliter
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Microgram/milliliter
  Day 1 | 0.417 (25.5) | 0.707 (44.7) | 0.888 (14.1)
  Day 3 | 0.398 (32.9) | 0.794 (35.7) | 1.080 (40.4)

44. Secondary Outcome: Tmax of GSK2982772 in Part B
Description: Blood samples were collected at indicated time points for analysis of Tmax
Time Frame: Pre-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 hours on Day 1 and Day 3
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Hours
  Day 1 | 4.058 [4.00 to 10.00] | 4.067 [4.00 to 12.00] | 4.000 [4.00 to 10.00]
  Day 3 | 4.000 [2.00 to 16.0] | 5.025 [4.00 to 20.00] | 4.000 [4.00 to 6.00]

45. Secondary Outcome: AUC (0-24) of GSK2982772 After Meal in Part C
Description: Blood samples were collected at indicated time points for analysis of AUC (0-24)
Time Frame: Pre-dose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram/milliliter
Groups:
- Part C MM-12h 480mg Delayed Fed (Standard): Participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fed state. Participants had received a dose before standard breakfast (delayed fed).
- Part C MM-12h 240mg Delayed Fed (High Fat): Participants received a single dose of 240 mg GSK2982772 MR MM-12hours (80% release at 12 hours). Participants had received a dose before high-fat breakfast (delayed fed).
- Part C MM-12h 480mg Fed (Standard): Participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fed state
Arm/Group | Part C MM-12h 480mg Delayed Fed (Standard) | Part C MM-12h 240mg Delayed Fed (High Fat) | Part C MM-12h 480mg Fed (Standard)
Number analyzed (Participants) | 15 | 14 | 16
Hours*microgram/milliliter | 17.505 (29.5) | 8.734 (47.4) | 21.543 (39.2)

46. Secondary Outcome: Cmax of GSK2982772 After Meal in Part C
Description: Blood samples were collected at indicated time points for analysis of Cmax
Time Frame: Pre-dose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/milliliter
Arm/Group | Part C MM-12h 480mg Delayed Fed (Standard) | Part C MM-12h 240mg Delayed Fed (High Fat) | Part C MM-12h 480mg Fed (Standard)
Number analyzed (Participants) | 15 | 14 | 16
Microgram/milliliter | 1.547 (40.8) | 1.064 (62.6) | 3.151 (32.5)

47. Secondary Outcome: C12 of GSK2982772 After Meal in Part C
Description: Blood samples were collected at indicated time points for analysis of C12
Time Frame: 12 hours post-dose
Population: PK Population. Only participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/milliliter
Arm/Group | Part C MM-12h 480mg Delayed Fed (Standard) | Part C MM-12h 240mg Delayed Fed (High Fat) | Part C MM-12h 480mg Fed (Standard)
Number analyzed (Participants) | 14 | 14 | 16
Microgram/milliliter | 0.706 (72.7) | 0.739 (37.1) | 0.317 (49.5)

48. Secondary Outcome: AUC(0-t) of GSK2982772 After Meal in Part C
Description: Blood samples were collected at indicated time points for analysis of AUC (0-t)
Time Frame: Pre-dose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram/milliliter
Arm/Group | Part C MM-12h 480mg Delayed Fed (Standard) | Part C MM-12h 240mg Delayed Fed (High Fat) | Part C MM-12h 480mg Fed (Standard)
Number analyzed (Participants) | 15 | 14 | 16
Hours*microgram/milliliter | 19.147 (28.0) | 9.202 (46.4) | 22.712 (36.2)

49. Secondary Outcome: AUC(0-inf) of GSK2982772 After Meal in Part C
Description: Blood samples were collected at indicated time points for analysis of AUC (0-inf) after meal.
Time Frame: Pre-dose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population. Only participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram/milliliter
Arm/Group | Part C MM-12h 480mg Delayed Fed (Standard) | Part C MM-12h 240mg Delayed Fed (High Fat) | Part C MM-12h 480mg Fed (Standard)
Number analyzed (Participants) | 7 | 6 | 5
Hours*microgram/milliliter | 18.941 (36.5) | 9.995 (62.4) | 24.367 (49.2)

50. Secondary Outcome: AUC(0-12) of GSK2982772 After Meal in Part C
Description: Blood samples were collected at indicated time points for analysis of AUC (0-12) after meal.
Time Frame: Pre-dose and at 2, 4, 6, 8, 10, and 12 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram/milliliter
Arm/Group | Part C MM-12h 480mg Delayed Fed (Standard) | Part C MM-12h 240mg Delayed Fed (High Fat) | Part C MM-12h 480mg Fed (Standard)
Number analyzed (Participants) | 15 | 14 | 16
Hours*microgram/milliliter | 17.111 (45.0) | 10.241 (45.9) | 6.771 (56.7)

51. Secondary Outcome: Frelformulation Based on AUC (0-t) of GSK2982772 After Meal in Part C
Description: Blood samples were collected at indicated time points for analysis of Frelformulation based on AUC of GSK2982772 after meal. Frel for Auc (0-t) was calculated as Geometric mean of AUC (0-t) of MM Fed formulation (fed) / Geometric mean of AUC (0-t) of MM Fasted Formulation (fasted) multiplied by 100.
Time Frame: Pre-dose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Groups:
- Part C:480mg MM-12hour Delayed Fed and 480 mg MM-12hour Fasted: Participants received single dose of 480 mg GSK2982772 MR MM-12hours (80% release at 12 hours) before standard breakfast (delayed fed) and received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fasted state. There was washout period of 7 days between doses
- Part C:480mg MM-12hour Fed and 480 mg MM- 12hour Fasted: Participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fed state and received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fasted state. There was washout period of 7 days between doses
- Part C:240mg MM-12hour Delayed Fed and 240mg MM-12hour Fasted: Participants received a single dose of 240 mg GSK2982772 MR MM-12hours (80% release at 12 hours) before high-fat breakfast (delayed fed)) and received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fasted state. There was washout period of 7 days between doses
Arm/Group | Part C:480mg MM-12hour Delayed Fed and 480 mg MM-12hour Fasted | Part C:480mg MM-12hour Fed and 480 mg MM- 12hour Fasted | Part C:240mg MM-12hour Delayed Fed and 240mg MM-12hour Fasted
Number analyzed (Participants) | 15 | 16 | 14
Percentage bioavailability | 94.69 [87.03 to 103.04] | 113.51 [104.52 to 123.27] | 91.13 [82.23 to 100.98]

52. Secondary Outcome: Frelformulation Based on Cmax of GSK2982772 After Meal in Part C
Description: Blood samples were collected at indicated time points for analysis of Frelformulation based on Cmax of GSK2982772 after meal. Frel for Cmax was calculated as Geometric mean of Cmax of MM Fed formulation (test) / Geometric mean of Cmax of MM Fasted Formulation (reference) multiplied by 100.
Time Frame: Pre-dose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Groups:
- Part C:240mg MM-12hour Delayed Fed and 240mg MM-12hour Fasted: Participants received a single dose of 240 mg GSK2982772 MR MM-12hours (80% release at 12 hours) before high-fat breakfast (delayed fed) and received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fasted state. There was washout period of 7 days between doses
Arm/Group | Part C:480mg MM-12hour Delayed Fed and 480 mg MM-12hour Fasted | Part C:480mg MM-12hour Fed and 480 mg MM- 12hour Fasted | Part C:240mg MM-12hour Delayed Fed and 240mg MM-12hour Fasted
Number analyzed (Participants) | 15 | 16 | 14
Percentage bioavailability | 76.56 [64.25 to 91.22] | 156.77 [132.06 to 186.09] | 113.81 [94.00 to 137.78]

53. Secondary Outcome: Tmax of GSK2982772 After Meal in Part C
Description: Blood samples were collected at indicated time points for analysis of Tmax of GSK2982772 after meal.
Time Frame: Pre-dose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 and 32 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C MM-12h 480mg Delayed Fed (Standard) | Part C MM-12h 240mg Delayed Fed (High Fat) | Part C MM-12h 480mg Fed (Standard)
Number analyzed (Participants) | 15 | 14 | 16
Hours | 4.000 [2.00 to 20.00] | 4.000 [2.00 to 10.02] | 5.017 [4.00 to 10.00]

54. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious AEs (SAE) in Part A
Description: An AE is any untoward medical occurrence in a clinical study participants, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly or birth defect and important medical events may jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed before. All participants who receive at least 1 dose of study treatment and were included in Safety Population. Participants will be analyzed according to the treatment they actually received.
Time Frame: Up to Day 43
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: IR 120mg Fasted | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 16 | 13 | 16
Participants
  Any AEs | 4 | 5 | 1 | 2
  Any SAEs | 0 | 1 | 0 | 0

55. Secondary Outcome: Number of Participants With AE and SAE in Part B
Description: An AE is any untoward medical occurrence in a clinical study participants, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly or birth defect and important medical events may jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Participants
  Any AEs | 1 | 3 | 1
  Any SAEs | 0 | 0 | 0

56. Secondary Outcome: Number of Participants With AE and SAE in Part C
Description: An AE is any untoward medical occurrence in a clinical study participants, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly or birth defect and important medical events may jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: Up to Day 43
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Part C:MM-12h 240mg Fasted: Participants received a single dose of 240 mg GSK2982772 MR MM-12hour tablet (80% release at 12 hours) in fasted state.
- Part C:MM-12h 480mg Fasted: Participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fasted state
- Part C:MM-12h 480mg Fed(Standard): Participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fed state
- Part C:MM-12h 480mg Delayed Fed(Standard): Participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fed state. Participants had received a dose before standard breakfast (delayed fed).
- Part C: MM-12h 240mg Delayed Fed(High Fat): Participants received a single dose of 240 mg GSK2982772 MR MM-12hours (80% release at 12 hours). Participants had received a dose before high-fat breakfast (delayed fed).
Arm/Group | Part C: IR 240mg Fasted | Part C:MM-12h 240mg Fasted | Part C:MM-12h 480mg Fasted | Part C:MM-12h 480mg Fed(Standard) | Part C:MM-12h 480mg Delayed Fed(Standard) | Part C: MM-12h 240mg Delayed Fed(High Fat)
Number analyzed (Participants) | 15 | 15 | 16 | 16 | 15 | 14
Participants
  Any AEs | 3 | 3 | 3 | 4 | 2 | 1
  Any SAEs | 0 | 0 | 0 | 0 | 0 | 0

57. Secondary Outcome: Number of Participants With Emergent Clinical Chemistry Results by Potential Clinical Importance Criteria: Part A
Description: Blood samples were collected for analysis of clinical chemistry parameters like albumin, creatinine, glucose, potassium, sodium, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), total bilirubin and calcium. Participants are counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants are counted twice if the subject has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Participants with missing Baseline value are assumed to have normal baseline value. Clinical chemistry parameters with potential clinical importance data has been reported. Data for worst-case post-Baseline has been reported.
Time Frame: Up to Day 43
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat) | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16 | 13 | 16 | 16
Participants
  ALT, low | 0 | 0 | 0 | 0
  ALT, normal or no change | 16 | 13 | 16 | 16
  ALT, high | 0 | 0 | 0 | 0
  Albumin, low | 0 | 0 | 0 | 0
  Albumin, normal or no change | 16 | 13 | 16 | 16
  Albumin, high | 0 | 0 | 0 | 0
  ALP, low | 0 | 0 | 0 | 0
  ALP, normal or no change | 16 | 13 | 16 | 16
  ALP, high | 0 | 0 | 0 | 0
  AST, low | 0 | 0 | 0 | 0
  AST, normal or no change | 16 | 13 | 16 | 16
  AST, high | 0 | 0 | 0 | 0
  Calcium, low | 0 | 0 | 0 | 0
  Calcium, normal or no change | 16 | 13 | 16 | 16
  Calcium, high | 0 | 0 | 0 | 0
  Creatinine, low | 0 | 0 | 0 | 0
  Creatinine, normal or no change | 16 | 13 | 16 | 16
  Creatinine, high | 0 | 0 | 0 | 0
  Glucose, low | 0 | 0 | 0 | 0
  Glucose, normal or no change | 16 | 13 | 16 | 16
  Glucose, high | 0 | 0 | 0 | 0
  Potassium, low | 0 | 0 | 0 | 0
  Potassium, normal or no change | 15 | 13 | 16 | 15
  Potassium, high | 1 | 0 | 0 | 1
  Sodium, low | 0 | 0 | 0 | 0
  Sodium, normal or no change16 | 16 | 13 | 16 | 16
  Sodium, high | 0 | 0 | 0 | 0
  Total Bilirubin, low | 0 | 0 | 0 | 0
  Total Bilirubin, normal or no change | 16 | 13 | 16 | 16
  Total Bilirubin, high | 0 | 0 | 0 | 0

58. Secondary Outcome: Number of Participants With Emergent Hematology Results by Potential Clinical Importance Criteria: Part A
Description: Blood samples were collected to analyze hematology parameters like platelet count, white blood cell (WBC) count, hemoglobin, hematocrit, total neutrophils, and lymphocytes. Participants are counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants are counted twice if the subject has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Participants with missing baseline value are assumed to have normal baseline value. Hematology parameters with potential clinical importance data has been reported. Data for worst-case post-Baseline has been reported.
Time Frame: Up to Day 43
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat) | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16 | 13 | 16 | 16
Participants
  Hematocrit, low | 0 | 0 | 0 | 0
  Hematocrit, normal or no change | 16 | 13 | 16 | 16
  Hematocrit, high | 0 | 0 | 0 | 0
  Hemoglobin, low | 0 | 0 | 0 | 0
  Hemoglobin, normal or no change | 16 | 13 | 16 | 16
  Hemoglobin, high | 0 | 0 | 0 | 0
  Lymphocytes, low | 0 | 0 | 0 | 0
  Lymphocytes, normal or no change | 16 | 13 | 16 | 16
  Lymphocytes, high | 0 | 0 | 0 | 0
  Platelet count, low | 0 | 0 | 0 | 0
  Platelet count, normal or no change | 16 | 13 | 16 | 16
  Platelet count, high | 0 | 0 | 0 | 0
  Total Neutrophils, low | 1 | 2 | 0 | 0
  Total Neutrophils, normal or no change | 15 | 11 | 16 | 16
  Total Neutrophils, high | 0 | 0 | 0 | 0
  WBC, low | 1 | 1 | 0 | 0
  WBC, normal or no change | 15 | 12 | 16 | 16
  WBC, high | 0 | 0 | 0 | 0

59. Secondary Outcome: Number of Participants Abnormal Urinalysis Dipstick Results: Part A
Description: Urine samples were collected for analysis of specific gravity, potential of hydrogen ions, glucose, protein, blood and ketones by dipstick method. Microscopic examination were performed if blood or protein values were abnormal.
Time Frame: Up to Day 43
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat) | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16 | 13 | 16 | 16
Participants | 0 | 0 | 0 | 0

60. Secondary Outcome: Number of Participants With Emergent Clinical Chemistry Results by Potential Clinical Importance Criteria: Part B
Description: Blood samples were collected for analysis of clinical chemistry parameters like albumin, creatinine, glucose, potassium, sodium, AST, ALT, ALP, total bilirubin and calcium. Participants are counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants are counted twice if the subject has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Participants with missing baseline value are assumed to have normal baseline value. Hematology parameters with potential clinical importance data has been reported. Data for worst-case post-Baseline has been reported.
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Participants
  ALT, low | 0 | 0 | 0
  ALT, normal or no change | 10 | 10 | 6
  ALT, high | 0 | 0 | 0
  Albumin, low | 0 | 0 | 0
  Albumin, normal or no change | 10 | 10 | 6
  Albumin, high | 0 | 0 | 0
  ALP, low | 0 | 0 | 0
  ALP, normal or no change | 10 | 10 | 6
  ALP, high | 0 | 0 | 0
  AST, low | 0 | 0 | 0
  AST, normal or no change | 10 | 10 | 6
  AST, high | 0 | 0 | 0
  Calcium, low | 0 | 0 | 0
  Calcium, normal or no change | 10 | 10 | 6
  Calcium, high | 0 | 0 | 0
  Creatinine, low | 0 | 0 | 0
  Creatinine, normal or no change | 10 | 10 | 6
  Creatinine, high | 0 | 0 | 0
  Glucose, low | 0 | 0 | 0
  Glucose, normal or no change | 10 | 10 | 6
  Glucose, high | 0 | 0 | 0
  Potassium, low | 0 | 0 | 0
  Potassium, normal or no change | 10 | 10 | 6
  Potassium, high | 0 | 0 | 0
  Sodium, low | 0 | 0 | 0
  Sodium, normal or no change | 10 | 10 | 6
  Sodium, high | 0 | 0 | 0
  Total Bilirubin, low | 0 | 0 | 0
  Total Bilirubin, normal or no change | 10 | 10 | 6
  Total Bilirubin, high | 0 | 0 | 0

61. Secondary Outcome: Number of Participants With Emergent Hematology Results by Potential Clinical Importance Criteria: Part B
Description: Blood samples were collected to analyze hematology parameters like platelet count, WBC count, hemoglobin, hematocrit, total neutrophils, and lymphocytes. Participants are counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants are counted twice if the subject has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Participants with missing baseline value are assumed to have normal baseline value. Hematology parameters with potential clinical importance data has been reported. Data for worst-case post-Baseline has been reported.
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Participants
  Hematocrit, low | 0 | 0 | 0
  Hematocrit, normal or no change | 10 | 10 | 6
  Hematocrit, high | 0 | 0 | 0
  Hemoglobin, low | 0 | 0 | 0
  Hemoglobin, normal or no change | 10 | 10 | 6
  Hemoglobin, high | 0 | 0 | 0
  Lymphocytes, low | 0 | 0 | 0
  Lymphocytes, normal or no change | 10 | 10 | 6
  Lymphocytes, high | 0 | 0 | 0
  Platelet count, low | 0 | 0 | 0
  Platelet count, normal or no change | 10 | 10 | 6
  Platelet count, high | 0 | 0 | 0
  Total Neutrophils, low | 0 | 0 | 0
  Total Neutrophils, normal or no change | 10 | 10 | 6
  Total Neutrophils, high | 0 | 0 | 0
  WBC, low | 0 | 0 | 0
  WBC, normal or no change | 10 | 10 | 6
  WBC, high | 0 | 0 | 0

62. Secondary Outcome: Number of Participants Abnormal Urinalysis Dipstick Results: Part B
Description: as for outcome 59
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Participants | 0 | 0 | 0

63. Secondary Outcome: Number of Participants With Emergent Clinical Chemistry Results by Potential Clinical Importance Criteria: Part C
Description: Blood samples were collected for analysis of clinical chemistry parameters like albumin, creatinine, glucose, potassium, sodium, AST, ALT, ALP, total bilirubin and calcium. Participants are counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants are counted twice if the participant has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Participants with missing Baseline value are assumed to have normal Baseline value. Clinical chemistry parameters with potential clinical importance data has been reported. Data for worst-case post-Baseline has been reported.
Time Frame: Up to Day 43
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: IR 240mg Fasted | Part C:MM-12h 240mg Fasted | Part C:MM-12h 480mg Fasted | Part C:MM-12h 480mg Fed(Standard) | Part C:MM-12h 480mg Delayed Fed(Standard) | Part C: MM-12h 240mg Delayed Fed(High Fat)
Number analyzed (Participants) | 15 | 15 | 16 | 16 | 15 | 14
Participants
  ALT, low | 0 | 0 | 0 | 0 | 0 | 0
  ALT, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  ALT, high | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, low | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  Albumin, high | 0 | 0 | 0 | 0 | 0 | 0
  ALP, low | 0 | 0 | 0 | 0 | 0 | 0
  ALP, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  ALP, high | 0 | 0 | 0 | 0 | 0 | 0
  AST, low | 0 | 0 | 0 | 0 | 0 | 0
  AST, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  AST, high | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, low | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  Calcium, high | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, low | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  Creatinine, high | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, low | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  Glucose, high | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, low | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  Potassium, high | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, low | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  Sodium, high | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, low | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, normal or no change | 15 | 15 | 15 | 16 | 14 | 14
  Total Bilirubin, high | 0 | 0 | 1 | 0 | 1 | 14

64. Secondary Outcome: Number of Participants With Emergent Hematology Results by Potential Clinical Importance Criteria: Part C
Description: Blood samples were collected to analyze hematology parameters like platelet count, WBC count, hemoglobin, hematocrit, total neutrophils, and lymphocytes. Participants are counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants are counted twice if the participant has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Participants with missing Baseline value are assumed to have normal Baseline value. Hematology parameters with potential clinical importance data has been reported. Data for worst-case post-Baseline has been reported.
Time Frame: Up to Day 43
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: IR 240mg Fasted | Part C:MM-12h 240mg Fasted | Part C:MM-12h 480mg Fasted | Part C:MM-12h 480mg Fed(Standard) | Part C:MM-12h 480mg Delayed Fed(Standard) | Part C: MM-12h 240mg Delayed Fed(High Fat)
Number analyzed (Participants) | 15 | 15 | 16 | 16 | 15 | 14
Participants
  Hematocrit, low | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  Hematocrit, high | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, low | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  Hemoglobin, high | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, low | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  Lymphocytes, high | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count, low | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  Platelet count, high | 0 | 0 | 0 | 0 | 0 | 0
  Total Neutrophils, low | 0 | 0 | 0 | 0 | 0 | 0
  Total Neutrophils, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  Total Neutrophils, high | 0 | 0 | 0 | 0 | 0 | 0
  WBC, low | 0 | 0 | 0 | 0 | 0 | 0
  WBC, normal or no change | 15 | 15 | 16 | 16 | 15 | 14
  WBC, high | 0 | 0 | 0 | 0 | 0 | 0

65. Secondary Outcome: Number of Participants Abnormal Urinalysis Dipstick Results: Part C
Description: as for outcome 59
Time Frame: Up to Day 43
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: IR 240mg Fasted | Part C:MM-12h 240mg Fasted | Part C:MM-12h 480mg Fasted | Part C:MM-12h 480mg Fed(Standard) | Part C:MM-12h 480mg Delayed Fed(Standard) | Part C: MM-12h 240mg Delayed Fed(High Fat)
Number analyzed (Participants) | 15 | 15 | 16 | 16 | 15 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0

66. Secondary Outcome: Number of Participants Abnormal Electrocardiogram (ECG) Findings: Part A
Description: Single 12-lead ECGs was obtained using an ECG machine. PR, QRS, QT and Corrected QT (QTc) intervals were measured in semi-supine or supine position. Number of participants with any visit post-Baseline abnormal clinically significant findings and abnormal not clinically significant findings in ECG results has been reported. Data for worst-case post-Baseline has been reported.
Time Frame: Up to Day 43
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat) | Part A: IR 120mg Fasted
Number analyzed (Participants) | 16 | 13 | 16 | 16
Participants
  Abnormal, not clinically significant | 6 | 8 | 9 | 9
  Abnormal, clinically significant | 1 | 0 | 0 | 0

67. Secondary Outcome: Number of Participants Abnormal ECG Findings: Part B
Description: Single 12-lead ECGs was obtained using an ECG machine. PR, QRS, QT and QTc intervals were measured in semi-supine or supine position. Number of participants with any visit post-Baseline abnormal clinically significant findings and abnormal not clinically significant findings in ECG results has been reported. Data for worst-case post-Baseline has been reported.
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Participants
  Abnormal, not clinically significant | 4 | 4 | 2
  Abnormal, clinically significant | 0 | 0 | 0

68. Secondary Outcome: Number of Participants Abnormal ECG Findings: Part C
Description: as for outcome 67
Time Frame: Up to Day 43
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: IR 240mg Fasted | Part C:MM-12h 240mg Fasted | Part C:MM-12h 480mg Fasted | Part C:MM-12h 480mg Fed(Standard) | Part C:MM-12h 480mg Delayed Fed(Standard) | Part C: MM-12h 240mg Delayed Fed(High Fat)
Number analyzed (Participants) | 15 | 15 | 16 | 16 | 15 | 14
Participants
  Abnormal, not clinically significant | 1 | 4 | 7 | 5 | 6 | 3
  Abnormal, clinically significant | 0 | 0 | 0 | 0 | 0 | 0

69. Secondary Outcome: Change From Baseline in Blood Pressure: Part A
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) was measured in semi-supine position. Baseline is defined as the latest pre-dose assessment before entering study. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24hours
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part A: IR 120mg Fasted | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 16 | 13 | 16
Millimeters of mercury
  SBP, Day 1, 2 hours, n=16,16, 13,16 | -1.4 (13.46) | 4.3 (10.70) | -0.2 (16.53) | -6.2 (11.20)
  SBP,Day 1, 12 hours, n=15,16, 13,16: number analyzed (Participants) | 15 | 16 | 13 | 16
  SBP,Day 1, 12 hours, n=15,16, 13,16 | -1.6 (14.05) | -2.5 (14.27) | -6.2 (12.34) | -2.9 (18.70)
  SBP,Day 2, 24 hours, n=16,16, 13,16 | 7.4 (13.86) | -2.7 (9.76) | -6.2 (11.22) | -3.9 (14.11)
  DBP, Day 1, 2 hours, n=16,16, 13,16 | 0.3 (7.33) | 3.0 (8.12) | -1.8 (7.81) | -4.4 (8.94)
  DBP,Day 1, 12 hours, n=16,16, 13,16 | -3.9 (10.01) | -3.6 (9.87) | -3.0 (9.27) | -3.9 (9.02)
  DBP,Day 2, 24 hours, n=16,16, 13,16 | 2.1 (8.51) | 0.7 (7.60) | -1.7 (7.79) | -1.1 (8.82)

70. Secondary Outcome: Change From Baseline in Heart Rate: Part A
Description: Heart rate was measured in semi-supine position. Baseline is defined as the latest pre-dose assessment before entering study. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 Pre-dose), Day 1: 2 and 12 hours; Day 2: 24hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A: IR 120mg Fasted | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 16 | 13 | 16
Beats per minute
  Day 1, 2 hours | -4.4 (5.11) | -0.3 (4.88) | -2.5 (7.62) | 3.9 (7.48)
  Day 1, 12 hours: number analyzed (Participants) | 15 | 16 | 13 | 16
  Day 1, 12 hours | 4.8 (6.06) | 5.2 (3.94) | 5.8 (5.57) | 7.5 (9.93)
  Day 2, 24 hours | 1.5 (9.41) | -2.1 (6.31) | 0.6 (7.14) | 0.9 (7.62)

71. Secondary Outcome: Change From Baseline in Respiration Rate: Part A
Description: Respiration rate was measured in semi-supine position. Baseline is defined as the latest pre-dose assessment before entering study. Change from Baseline was defined as post-dose visit value minus Baseline value
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part A: IR 120mg Fasted | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 16 | 13 | 16
Breaths per minute
  Day 1, 2 hours | -0.4 (1.67) | 0.8 (1.65) | 0.0 (1.00) | -1.5 (2.50)
  Day 1, 12 hours: number analyzed (Participants) | 15 | 16 | 13 | 16
  Day 1, 12 hours | -0.6 (1.71) | -0.1 (1.82) | -0.2 (1.21) | -2.4 (2.63)
  Day 2, 24 hours | 1.3 (2.15) | -0.1 (1.54) | -1.5 (1.51) | -1.4 (2.13)

72. Secondary Outcome: Change From Baseline in Body Temperature: Part A
Description: Body temperature was measured in semi-supine position. Baseline is defined as the latest pre-dose assessment before entering study. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part A: IR 120mg Fasted | Part A: MT-12hour 120mg Fasted | Part A: MT-8hour 120mg Fasted | Part A: MT-12hour 120mg Fed (High Fat)
Number analyzed (Participants) | 16 | 16 | 13 | 16
Degree Celsius
  Day 1, 2 hours | 0.02 (0.152) | 0.18 (0.180) | 0.05 (0.145) | 0.14 (0.126)
  Day 1, 12 hours: number analyzed (Participants) | 15 | 16 | 13 | 16
  Day 1, 12 hours | 0.07 (0.139) | -0.04 (0.145) | 0.13 (0.118) | 0.11 (0.173)
  Day 2, 24 hours | 0.04 (0.182) | 0.07 (0.095) | 0.12 (0.114) | 0.12 (0.161)

73. Secondary Outcome: Change From Baseline in Blood Pressure: Part B
Description: SBP and DBP was measured in semi-supine position. Baseline is defined as the latest pre-dose assessment before entering study. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 1 and Day 3: 2 and 12 hours; Pre-dose on Days 2 and 3; Day 4: 24 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Millimeters of mercury
  SBP, Day 1, 2 hours | -0.5 (7.40) | 5.4 (7.37) | 1.2 (7.08)
  SBP,Day 1, 12 hours | 2.7 (7.75) | 1.5 (8.86) | 1.0 (10.73)
  SBP,Day 2, Pre-dose | -0.1 (5.26) | 3.5 (7.76) | 1.8 (6.62)
  SBP,Day 3, Pre-dose | -1.0 (9.35) | 1.1 (5.09) | -0.7 (14.09)
  SBP,Day 3, 2 hours | 2.0 (8.37) | 5.5 (9.51) | -3.3 (9.14)
  SBP,Day 3, 12 hours | 2.4 (11.55) | 7.4 (14.17) | 3.8 (8.21)
  SBP,Day 4, 24 hours | 2.9 (9.22) | 6.1 (5.04) | 6.0 (11.24)
  DBP, Day 1, 2 hours | 2.4 (7.31) | 2.1 (7.16) | -4.0 (4.20)
  DBP,Day 1, 12 hours | -1.7 (5.50) | -2.2 (4.59) | -5.7 (4.03)
  DBP,Day 2, Pre-dose | -1.5 (4.55) | 2.0 (7.47) | -2.7 (6.56)
  DBP,Day 3, Pre-dose | 2.6 (8.57) | 1.3 (6.65) | 1.3 (4.50)
  DBP,Day 3, 2 hours | 3.1 (7.00) | 4.0 (5.31) | -5.8 (3.87)
  DBP,Day 3, 12 hours | -1.4 (7.78) | -1.4 (5.72) | -2.5 (2.81)
  DBP,Day 4, 24 hours | 3.0 (5.56) | 4.6 (4.77) | 1.3 (6.65)

74. Secondary Outcome: Change From Baseline in Heart Rate: Part B
Description: as for outcome 70
Time Frame: Baseline (Day 1, Pre-dose), Day 1 and Day 3: 2 and 12 hours; Pre-dose on Days 2 and 3; Day 4: 24 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Beats per minute
  Day 1, 2 hours | 0.0 (5.50) | -2.4 (5.38) | 7.3 (6.89)
  Day 1, 12 hours | 10.0 (4.00) | 8.8 (5.22) | 10.5 (3.78)
  Day 2, Pre-dose | -0.1 (4.68) | -0.8 (6.37) | -1.8 (2.71)
  Day 3, Pre-dose | 2.3 (4.74) | -0.1 (5.88) | 1.5 (5.43)
  Day 3, 2 hours | 1.2 (5.37) | -0.3 (5.36) | 4.0 (2.28)
  Day 3, 12 hours | 8.6 (4.58) | 10.6 (7.26) | 7.7 (5.28)
  Day 4, 24 hours | 4.7 (8.64) | 6.7 (10.01) | 0.3 (2.58)

75. Secondary Outcome: Change From Baseline in Respiration Rate: Part B
Description: as for outcome 71
Time Frame: Baseline (Day 1, Pre-dose), Day 1 and Day 3: 2 and 12 hours; Pre-dose on Days 2 and 3; Day 4 24 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Breaths per minute
  Day 1, 2 hours | 0.5 (2.27) | -2.0 (2.00) | -1.2 (3.54)
  Day 1, 12 hours | -0.1 (1.37) | -2.5 (2.17) | -1.5 (2.35)
  Day 2, Pre-dose | -0.3 (1.49) | -0.5 (2.07) | -0.5 (2.74)
  Day 3, Pre-dose | -0.7 (2.67) | -0.5 (1.43) | 1.5 (2.26)
  Day 3, 2 hours | -1.3 (2.36) | -1.0 (2.21) | -0.7 (2.16)
  Day 3, 12 hours | 0.3 (3.02) | -1.3 (2.16) | -0.8 (1.33)
  Day 4, 24 hours | -0.8 (1.87) | -1.0 (1.89) | -0.3 (2.42)

76. Secondary Outcome: Change From Baseline in Body Temperature: Part B
Description: as for outcome 72
Time Frame: Baseline (Day 1, Pre-dose), Day 1 and Day 3: 2 and 12 hours; Pre-dose on Days 2 and 3; Day 4: 24 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part B: MT-12 120mg Fasted | Part B :MT-12 240mg Fasted | Part B :MT-12hour 300mg Fed (Standard)
Number analyzed (Participants) | 10 | 10 | 6
Degree Celsius
  Day 1, 2 hours | 0.03 (0.298) | -0.01 (0.233) | 0.00 (0.110)
  Day 1, 12 hours | 0.06 (0.181) | 0.08 (0.274) | 0.07 (0.082)
  Day 2, Pre-dose | 0.04 (0.184) | -0.04 (0.158) | 0.12 (0.133)
  Day 3, Pre-dose | 0.04 (0.135) | 0.07 (0.271) | 0.23 (0.151)
  Day 3, 2 hours | -0.03 (0.149) | 0.01 (0.260) | -0.08 (0.147)
  Day 3, 12 hours | 0.01 (0.191) | 0.05 (0.242) | 0.05 (0.138)
  Day 4, 24 hours | 0.04 (0.171) | 0.11 (0.247) | 0.00 (0.089)

77. Secondary Outcome: Change From Baseline in Blood Pressure: Part C
Description: as for outcome 73
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part C: IR 240mg Fasted | Part C:MM-12h 240mg Fasted | Part C:MM-12h 480mg Fasted | Part C:MM-12h 480mg Fed(Standard) | Part C:MM-12h 480mg Delayed Fed(Standard) | Part C: MM-12h 240mg Delayed Fed(High Fat)
Number analyzed (Participants) | 15 | 15 | 16 | 16 | 15 | 14
Millimeters of mercury
  SBP, Day 1, 2 hours | -3.3 (7.93) | -0.6 (7.50) | -0.6 (6.16) | -4.9 (9.18) | 1.1 (16.02) | -0.2 (11.44)
  SBP,Day1, 12 hours | -3.1 (10.04) | -2.6 (8.34) | 1.4 (12.06) | 0.1 (10.81) | -7.3 (14.92) | 0.9 (16.03)
  SBP,Day2, 24 hours | 4.9 (8.02) | -1.4 (6.71) | -1.6 (8.39) | -3.1 (8.50) | 2.6 (10.84) | -7.5 (10.58)
  DBP, Day 1, 2 hours | -0.1 (7.41) | -0.7 (6.43) | 2.0 (6.92) | -4.3 (6.94) | -0.6 (7.88) | -1.9 (5.50)
  DBP,Day1, 12 hours | -2.1 (7.23) | -1.1 (6.36) | -3.1 (6.53) | -0.6 (8.02) | -3.7 (9.61) | 0.0 (8.38)
  DBP,Day2, 24 hours | 0.4 (7.21) | 1.0 (4.88) | -0.5 (6.64) | 2.8 (6.37) | 0.7 (7.49) | 2.4 (6.21)

78. Secondary Outcome: Change From Baseline in Heart Rate: Part C
Description: as for outcome 70
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part C: IR 240mg Fasted | Part C:MM-12h 240mg Fasted | Part C:MM-12h 480mg Fasted | Part C:MM-12h 480mg Fed(Standard) | Part C:MM-12h 480mg Delayed Fed(Standard) | Part C: MM-12h 240mg Delayed Fed(High Fat)
Number analyzed (Participants) | 15 | 15 | 16 | 16 | 15 | 14
Beats per minute
  Day 1, 2 hours | 2.1 (6.94) | -5.3 (6.19) | 0.0 (6.86) | 7.3 (6.56) | 8.2 (5.72) | 8.2 (7.32)
  Day 1, 12 hours | 6.8 (6.20) | 6.5 (9.73) | 11.2 (9.65) | 10.3 (6.94) | 9.3 (8.28) | 8.6 (6.99)
  Day 2, 24 hours | 1.8 (5.44) | 0.1 (6.41) | -0.4 (3.77) | 0.4 (5.80) | -0.9 (6.19) | 1.6 (7.74)

79. Secondary Outcome: Change From Baseline in Respiration Rate: Part C
Description: as for outcome 71
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part C: IR 240mg Fasted | Part C:MM-12h 240mg Fasted | Part C:MM-12h 480mg Fasted | Part C:MM-12h 480mg Fed(Standard) | Part C:MM-12h 480mg Delayed Fed(Standard) | Part C: MM-12h 240mg Delayed Fed(High Fat)
Number analyzed (Participants) | 15 | 15 | 16 | 16 | 15 | 14
Breaths per minute
  Day 1, 2 hours | 1.7 (3.37) | 0.6 (2.03) | 0.9 (2.90) | -1.1 (2.95) | 1.8 (1.74) | 0.1 (2.76)
  Day 1, 12 hours | 1.1 (2.59) | 1.0 (2.85) | 0.6 (2.66) | -1.1 (2.90) | -0.3 (2.61) | 0.5 (1.51)
  Day 2, 24 hours | 1.6 (3.25) | 0.4 (3.07) | 0.6 (4.00) | -2.2 (2.66) | 1.8 (2.31) | 0.4 (3.34)

80. Secondary Outcome: Change From Baseline in Body Temperature: Part C
Description: as for outcome 72
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part C: IR 240mg Fasted | Part C:MM-12h 240mg Fasted | Part C:MM-12h 480mg Fasted | Part C:MM-12h 480mg Fed(Standard) | Part C:MM-12h 480mg Delayed Fed(Standard) | Part C: MM-12h 240mg Delayed Fed(High Fat)
Number analyzed (Participants) | 15 | 15 | 16 | 16 | 15 | 14
Degree Celsius
  Day 1, 2 hours | -0.10 (0.245) | -0.05 (0.192) | -0.07 (0.215) | 0.23 (0.275) | 0.01 (0.228) | 0.10 (0.301)
  Day 1, 12 hours | 0.02 (0.197) | -0.11 (0.229) | -0.05 (0.271) | 0.12 (0.307) | -0.14 (0.241) | -0.10 (0.266)
  Day 2, 24 hours | -0.04 (0.256) | 0.15 (0.261) | -0.00 (0.239) | 0.10 (0.278) | -0.09 (0.269) | -0.01 (0.241)

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected up to Day 43 for Part A and Part C and up to Day 22 for Part B
Description: Non-serious AEs and SAEs were collected in Safety population.
Groups:
- Part A:IR 120mg Fasted: Participants received a single oral dose of 120 mg GSK2982772 (4x30 mg) IR tablet in fasted state
- Part A:MT-12hour 120mg Fed (High Fat): Participants received single oral dose of 120 mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) after high fat meal
- Part B:MT-12hour 120mg Fasted: Participants received once daily dose of 120mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fasted state for 3 days.
- Part B:MT-12hour 240mg Fasted: Participants received once daily dose of 240mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fasted state for 3 days
- Part B:MT-12hour 300mg Fed (Standard): Participants received once daily dose of 300mg GSK2982772 MR MT-12hour capsule (80% release at 12 hours) in fed state (standard meal) for 3 days
- Part C:IR 240mg Fasted: Participants received a single dose of 240 mg GSK2982772 IR tablet in fasted state
- Part C:MM-12hour 240mg Fasted: Participants received a single dose of 240 mg GSK2982772 MR MM-12hour tablet (80% release at 12 hours) in fasted state
- Part C:MM-12hour 480mg Fasted: Participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fasted state
- Part C:MM-12hour 480mg Fed (Standard): Participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fed state
- Part C:MM-12hour 480mg Delayed Fed (Standard): Participants received a single dose of 480 mg GSK2982772 MR MM-12 hour tablet (80% release at 12 hours) in fed state. Participants had received a dose before standard breakfast (delayed fed).
- Part C:MM-12hour 240mg Delayed Fed (High Fat): Participants received a single dose of 240 mg GSK2982772 MR MM-12hours (80% release at 12 hours). Participants had received a dose before high-fat breakfast (delayed fed).
Arm/Group | Part A:IR 120mg Fasted | Part A:MT-12hour 120mg Fasted | Part A:MT-8hour 120mg Fasted | Part A:MT-12hour 120mg Fed (High Fat) | Part B:MT-12hour 120mg Fasted | Part B:MT-12hour 240mg Fasted | Part B:MT-12hour 300mg Fed (Standard) | Part C:IR 240mg Fasted | Part C:MM-12hour 240mg Fasted | Part C:MM-12hour 480mg Fasted | Part C:MM-12hour 480mg Fed (Standard) | Part C:MM-12hour 480mg Delayed Fed (Standard) | Part C:MM-12hour 240mg Delayed Fed (High Fat)
All-Cause Mortality (participants affected / at risk) | 0/16 | 1/16 | 0/13 | 0/16 | 0/10 | 0/10 | 0/6 | 0/15 | 0/15 | 0/16 | 0/16 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/16 | 0/13 | 0/16 | 0/10 | 0/10 | 0/6 | 0/15 | 0/15 | 0/16 | 0/16 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 4/16 | 5/16 | 1/13 | 2/16 | 1/10 | 3/10 | 1/6 | 3/15 | 3/15 | 3/16 | 4/16 | 2/15 | 1/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A:IR 120mg Fasted (N=16) | Part A:MT-12hour 120mg Fasted (N=16) | Part A:MT-8hour 120mg Fasted (N=13) | Part A:MT-12hour 120mg Fed (High Fat) (N=16) | Part B:MT-12hour 120mg Fasted (N=10) | Part B:MT-12hour 240mg Fasted (N=10) | Part B:MT-12hour 300mg Fed (Standard) (N=6) | Part C:IR 240mg Fasted (N=15) | Part C:MM-12hour 240mg Fasted (N=15) | Part C:MM-12hour 480mg Fasted (N=16) | Part C:MM-12hour 480mg Fed (Standard) (N=16) | Part C:MM-12hour 480mg Delayed Fed (Standard) (N=15) | Part C:MM-12hour 240mg Delayed Fed (High Fat) (N=14)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A:IR 120mg Fasted (N=16) | Part A:MT-12hour 120mg Fasted (N=16) | Part A:MT-8hour 120mg Fasted (N=13) | Part A:MT-12hour 120mg Fed (High Fat) (N=16) | Part B:MT-12hour 120mg Fasted (N=10) | Part B:MT-12hour 240mg Fasted (N=10) | Part B:MT-12hour 300mg Fed (Standard) (N=6) | Part C:IR 240mg Fasted (N=15) | Part C:MM-12hour 240mg Fasted (N=15) | Part C:MM-12hour 480mg Fasted (N=16) | Part C:MM-12hour 480mg Fed (Standard) (N=16) | Part C:MM-12hour 480mg Delayed Fed (Standard) (N=15) | Part C:MM-12hour 240mg Delayed Fed (High Fat) (N=14)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye haematoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injury associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03266172/Prot_001.pdf
  • Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT03266172/SAP_000.pdf